CLINICAL TRIAL: NCT03476811
Title: Postoperative subQ Pain Control for Spinal Fusion Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Robert Bina, Neurosurgery Resident, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1712090332
Record Dates: First submitted 2018-02-22; First posted 2018-03-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Spine Fusion; Surgery; Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: This trial is a comparative trial investigating outcomes in 3 parallel groups. The control group will receive standard of care pain control following surgery, the Marcaine group will receive infusion of FDA approved Marcaine around the operative site following surgery through an FDA approved surgical device. The Placebo group will have the drug delivery device implanted with delivery of saline.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Control Group (No Intervention): Normal treatment paradigm (no anesthetic pump) with pain medications, only.
- Marciano Group (Active Comparator): Subcutaneous pain control with OnQ pump (0.25% Marcaine at 2ml/hr) and pain medications.
  Interventions: Drug: 0.25% Marcaine at 2ml/hr and pain medications
- Placebo Group (Placebo Comparator): OnQ pump with placebo (normal saline at 2ml/hr) and pain medications.
  Interventions: Device: Placement of OnQ Drug pump

INTERVENTIONS:
Drug: 0.25% Marcaine at 2ml/hr and pain medications — Subcutaneous pain control with OnQ Subcutaneous Drug pump
  Other Names: OnQ Subcutaneous Drug pump
  Arms: Marciano Group
Device: Placement of OnQ Drug pump — Subcutaneous placement of OnQ drug pump with normal saline infusion
  Arms: Placebo Group

SUMMARY:
Post-operative pain following lumbar spine fusion is frequently difficult to manage and can lead to increased doses of opiate pain medications to control pain. In this study, the use of subcutaneous local anesthesia will be studied to determine its efficacy at reducing post-operative pain following spinal fusion surgery.

DETAILED DESCRIPTION:
For patients randomized to the experimental or to the placebo groups, two subcutaneous catheters will be tunneled under the skin with large hollow-bore needles along the entire length of the incision on either side prior to closure. These catheters will deliver study drug (0.25% Marcaine) directly into the incision. They will be affixed to the skin with steri-strips. The catheters will then be attached to a drug delivery pump at 2mL/hour and will be removed prior to discharge.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years of age or greater
* Surgery to be done at Banner University Medical Center-Tucson
* Elective Surgeries only
* Lower Thoracic or Lumbar fusions only - Posterior Approach
* Postero or Posterolateral Instrumented Fusions with or without Interbody graft
* Transforaminal Interbody Fusions
* Must be able to cooperate in the daily VAS assessment

Exclusion Criteria:

* Patients under 18 years of age
* Prisoners
* Pregnant women
* Hypersensitivity to infusion medication
* Deformity Correction cases requiring osteotomies
* Surgical fusion in acute phase for traumatic injury
* Anterior Lumbar Interbody Fusion, Direct Lateral Interbody Fusion procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-02-09 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Pain control | From post operative day 1 until patient discharge or 30 days, whichever comes first
  A daily Visual Analog Score Pain scale (1-10) for pain severity, (1 least pain, 10 most pain) will be assessed and recorded daily by a blinded assessor.

SECONDARY OUTCOMES:
Time to discharge | from the day of hospital admission to the day of hospital discharge or 45 days, whichever comes first.
  Number of hospital days from time when patient surgery is completed to discharge will be assessed
Total Milligrams of IV pain medication | from the first post-operative dose of IV pain medication until the last dose prior to discharge from the hospital or 45 days, whichever comes first
  Total milligrams of IV pain medications will be assessed
Total Doses of IV pain medication | from the first post-operative dose of IV pain medication until the last dose prior to discharge from the hospital or 45 days, whichever comes first
  Number of doses of IV pain medications will be assessed
Total Milligrams of oral pain medication | from the first post-operative dose of oral pain medication until the last dose prior to discharge from the hospital or 45 days, whichever comes first
  Total milligrams of oral pain medications will be assessed
Total Doses of oral pain medication | from the first post-operative dose of oral pain medication until the last dose prior to discharge from the hospital or 45 days, whichever comes first
  Total doses of oral pain medications will be assessed

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gottschalk A, Freitag M, Tank S, Burmeister MA, Kreil S, Kothe R, Hansen-Algenstedt N, Weisner L, Staude HJ, Standl T. Quality of postoperative pain using an intraoperatively placed epidural catheter after major lumbar spinal surgery. Anesthesiology. 2004 Jul;101(1):175-80. doi: 10.1097/00000542-200407000-00027. PMID 15220788
- [Background] Perkins FM, Kehlet H. Chronic pain as an outcome of surgery. A review of predictive factors. Anesthesiology. 2000 Oct;93(4):1123-33. doi: 10.1097/00000542-200010000-00038. No abstract available. PMID 11020770
- [Background] Manchikanti L, Singh V, Cash KA, Pampati V, Datta S. Management of pain of post lumbar surgery syndrome: one-year results of a randomized, double-blind, active controlled trial of fluoroscopic caudal epidural injections. Pain Physician. 2010 Nov-Dec;13(6):509-21. PMID 21102963
- [Background] Reynolds RA, Legakis JE, Tweedie J, Chung Y, Ren EJ, Bevier PA, Thomas RL, Thomas ST. Postoperative pain management after spinal fusion surgery: an analysis of the efficacy of continuous infusion of local anesthetics. Global Spine J. 2013 Mar;3(1):7-14. doi: 10.1055/s-0033-1337119. Epub 2013 Mar 2. PMID 24436846